CLINICAL TRIAL: NCT01580878
Title: A Double-Blind, Randomized, Parallel-Group, Vehicle-Controlled, Multicenter Study to Evaluate the Safety and Bioequivalence of a Generic Butenafine Hydrochloride Cream, 1% and Reference Listed Lotrimin Ultra® (Butenafine Hydrochloride Cream, 1%) and Compare Both Active Treatments to a Vehicle Control in the Treatment of Interdigital Tinea Pedis.
Brief Title: Evaluate the Safety & Bioequivalence of a Generic Butenafine Cream & Lotrimin Ultra® & Compare Both to a Vehicle Control in Treatment of Interdigital Tinea Pedis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTNF 1104
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Tinea Pedis
Keywords: Butenafine Hydrochloride Cream, 1%; Lotrimin Ultra® Cream, 1%; Interdigital Tinea Pedis; Safety and Bioequivalence
MeSH Terms: conditions — Tinea Pedis | interventions — butenafine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Butenafine Hydrochloride Cream, 1% (Experimental): Butenafine Hydrochloride Cream, 1% (Taro Pharmaceuticals, Inc.)
  Interventions: Drug: Butenafine Hydrochloride Cream, 1%
- Lotrimin Ultra® (Active Comparator): Lotrimin Ultra® (Butenafine Hydrochloride Cream, 1%) (Schering Plough HealthCare Products Inc.)
  Interventions: Drug: Lotrimin Ultra®
- Butenafine Vehicle (Placebo Comparator): Butenafine Cream vehicle (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Butenafine Vehicle

INTERVENTIONS:
Drug: Butenafine Hydrochloride Cream, 1% — Butenafine Hydrochloride Cream, 1% applied twice daily for 7 consecutive days
  Arms: Butenafine Hydrochloride Cream, 1%
Drug: Lotrimin Ultra® — Lotrimin Ultra® (Butenafine Hydrochloride Cream, 1%) applied twice daily for 7 consecutive days.
  Arms: Lotrimin Ultra®
Drug: Butenafine Vehicle — Butenafine Vehicle applied twice daily for 7 consecutive days.
  Arms: Butenafine Vehicle

SUMMARY:
The primary objective of this study is to determine the comparability of the safety and efficacy of a generic Butenafine Hydrochloride Cream, 1% (test product) and Lotrimin Ultra® (the reference listed drug) in subjects with interdigital tinea pedis. It will also be determined whether the efficacy of each of the two active treatments is superior to that of the vehicle cream (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Willing & able to provide & understand written informed consent
* Healthy male or non-pregnant, non-lactating female at least 18 years of age and older
* Clinical diagnosis of tinea pedis with lesions localized to the interdigital spaces or that is predominantly interdigital but may extend to other areas
* Tinea pedis provisionally confirmed at baseline by positive potassium hydroxide (KOH)wet mount preparation showing segmented fungal hyphae
* Has sum of the clinical signs and symptoms scores of the target lesion of at least 4, including a minimum score of 2 for erythema & a minimum score of 2 for scaling or pruritus
* Currently in general good health with no clinically significant disease
* Willing and able to understand and comply with study requirements
* Women of childbearing potential must have a negative urine pregnancy test and be willing to use an acceptable form of birth control during study

Exclusion Criteria:

* Females who are pregnant, breastfeeding, planning a pregnancy, or do not agree to use an acceptable form of birth control during the study
* Confluent, diffuse moccasin-type tinea pedis of the entire plantar surface
* Presence of any other infection of the foot or other disease that might confound treatment evaluation
* History of dermatophyte infections unresponsive to antifungal drugs
* Known hypersensitivity to Butenafine Hydrochloride or any component of the study medications
* Use of antipruritics, topical systemic corticosteroid, antibiotic or antifungal therapy, oral terbinafine or itraconazole, or immunosuppressive medication or radiation therapy more recently than indicated washout period
* Current oral, vaginal, or mucocutaneous candidiasis
* Current bacterial skin infection, secondary cellulitis, lymphangitis, or pyoderma
* Presence of current conditions that require systemic antimicrobial or antifungal therapy
* Uncontrolled diabetes mellitus, peripheral vascular disease, chronic venous stasis, or other significant condition
* Current severe onychomycosis
* Any clinically significant condition or situation, other than condition being studied, that would interfere with the study evaluations or participation
* Use of any investigational drugs or device within 30 days of signing Informed Consent Form (ICF)
* Current participation in any other clinical study
* Consumes excessive amounts of alcohol, abuses drugs, or has any condition that would compromise compliance
* Previous participation in this study
* Subjects with past history of tinea pedis with lack of response to antifungal therapy
* Subjects who in Investigator's opinion would be non-compliant
* Employees or direct relatives of an employee of the study center or Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Therapeutic Cure | 42 days
  Subjects with both clinical cure and mycologic cure are considered therapeutic cures.

CONTACTS AND LOCATIONS:
Overall Officials: Symbio CRO, Study Chair — http://symbioresearch.com/